CLINICAL TRIAL: NCT02695134
Title: Healing Touch Intervention in Post-Cardiac Event Patients Prior to Starting a Cardiac Rehab Program
Brief Title: Healing Touch Prior to Cardiac Rehab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scripps Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB-16-6754
Record Dates: First submitted 2016-02-23; First posted 2016-03-01 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Heart Disease
MeSH Terms: conditions — Heart Diseases | interventions — Touch

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Other): This group will receive 6 Healing Touch treatments over 3 weeks
  Interventions: Other: Healing Touch
- Control Group[ (No Intervention): This group will continue with their usual medical treatments but receive NO Healing Touch

INTERVENTIONS:
Other: Healing Touch — Healing Touch (HT) is an energy based approach to health and healing. It uses light touch to influence the energy field that surrounds the body, and energy centers which control the flow of energy to the physical body.
  Arms: Intervention Group

SUMMARY:
The purpose of the investigators proposed randomized, controlled study is to examine the effect of 6 one hour treatments of Healing Touch (HT) over 3 weeks on post-cardiac event patients, while they wait to enter a Cardiac Rehab (CR) program.Patients enrolled in the Scripps Center for Integrative Medicine (SCIM) Cardiac Rehab Program typically experience a waiting period of 3 weeks, or sometimes more, before starting the program.

Secondary aims of the proposed study are to evaluate the effect of HT on CR program outcome measures of METs, BMI, physical and mental well-being, and attendance in this population.

New participants in the CR program who qualify and agree to participate in the study will be consented and randomly assigned to the Intervention Group who will receive Healing Touch therapy, or to the Control Group, which will not receive HT.

At baseline both groups will complete the Dartmouth Quality of Life and SF-36 Health Surveys. The questionnaires will be repeated at the end of the 3 week study period and at the end of the 3 months SCIM CR program.

An effect size of 15% was chosen, with an alpha level of 0.05, 80% power, 95% confidence level, and using a two-tailed test, it was determined that a sample size of 56 patients in each group would be needed for between group comparisons. To account for potential attrition the study will enroll 124 subjects, 62 in each group.

Our rationale is that Healing Touch, in addition to standard medical care will reduce post-cardiac event stress and anxiety symptoms in patients waiting to enter a cardiac rehab program, as measured by the Dartmouth Quality of Life Index and the SF36 questionnaire. Further, the investigators suggest that Healing Touch treatments will improve patient's final outcomes of the 12 week CR program.

DETAILED DESCRIPTION:
Study Plan

HEALING TOUCH Healing Touch (HT) is an energy based approach to health and healing. It uses light touch to influence the energy field that surrounds the body, and energy centers which control the flow of energy to the physical body. HT can restore harmony and balance, which can affect all physical, mental, emotional, and spiritual health, as well as self-healing. HT complements traditional health care and is used together with other approaches to health and healing.

Healing touch has been studied for use in pain, cancer, endocrine-immune-HIV, mental health, and cardiovascular factors in patients ranging from pediatric to the elderly.

POST-CARDIAC EVENT STRESS AND ANXIETY SYMPTOMS Having a major cardiac event can be a stressful, life changing occurrence. Often, the psychological impacts of having a heart attack (myocardial infarction) are underestimated and can be long lasting. In fact, there is evidence to suggest that the emotional stressors that occur post-MI are consistent with symptoms of post-traumatic stress disorder (PTSD), which has been shown to be associated with higher rates of recurrent coronary events and overall increased mortality in diagnosed patients.

Studies have shown that mental stress has a negative effect on a person's heart health. In particular:

* Unmanaged stress can lead to high blood pressure, arterial damage, irregular heart rhythms and a weakened immune system.
* Patients with depression have been shown to have increased platelet reactivity, decreased heart variability and increased pro-inflammatory markers (such as C-reactive protein or CRP), which are all risk factors for cardiovascular disease.
* For people with heart disease, depression can increase the risk of an adverse cardiac event such as a heart attack or blood clots. For people who do not have heart disease, depression can also increase the risk of a heart attack and development of coronary artery disease.
* In one landmark study, the continued presence of depression after recovery increased the risk of death (mortality) to 17 percent within 6 months after a heart attack (versus 3 percent mortality in heart attack patients who didn't have depression). Frasure-Smith N, et al. Depression following myocardial infarction: Impact on 6-month survival. JAMA, October 20, 1993. 270(15):1819-1825.

RELATED STUDIES

HEALING TOUCH has been in use at Scripps hospitals since 1993. The Cardiac Healing Touch Program at the Scripps Center for Integrative Medicine at Scripps Clinic and Scripps Green Hospital collected data on 305 cardiac surgery patients. Unpublished outcomes revealed that post-surgical cardiac patients experienced a 74% reduction in pain and a 71% reduction in anxiety after receiving HT.

In another study performed by the Scripps Center for Integrative Medicine at a Marine Base near San Diego, called Complementary Medicine for PTSD and Related Symptoms in Returning Active Duty Military, revealed statistically and clinically significant reduction in PTSD (p <.0005, Cohen's d = .85), as well as depression (p <.0005, Cohen's d = .70) for the healing touch and guided imagery intervention versus the control group.

Post-cardiac event patients who have been referred to a Cardiac Rehab program often find that they are being asked to wait before a position becomes available in the CR program. In some programs this may involve a waiting period of several weeks. At the Scripps Center for Integrative Medicine Cardia Rehab program the waiting period is typically 3 weeks, or slighly more. During this period, many patients find that their stress and anxiety levels in reaction to their recent cardiac event remain untreated. It is this group of patients the investigators aim to enroll into the research study to determine whether 6 healing touch treatments during a waiting period of 3 weeks will decrease their stress and anxiety before entering the cardiac rehab program. Moreover, the investigators will follow the patients through CR and determine whether the pre-program HT treatments improve the patient's overall physical outcomes measures.

Research Methods

Baseline Assessment Upon enrollment in the study, including signing the consent, participants will answer questionnaires to assess their baseline status including demographics, brief medical history, and the following two questionnaires: Dartmouth Quality of Life and SF-36 Health Survey.

Randomization Following initial assessment, participants will be randomly assigned to the Intervention Group who will receive Healing Touch therapy, or to the Control Group, which will not receive HT. All study participants will enter the CR program after either 3 weeks of HT intervention or a 3 week waiting period. If there is no opening available immediately following the 3 week period, study subjects will be entered into the program as soon as a space is available.

Intervention Group

The HT group will receive two one hour sessions per week for a total of 6 sessions, over 3 weeks. Healing Touch practitioners who have completed the healing touch program and are certified healing touch practitioners will perform the healing touch sessions. Whenever possible each patient will be given the treatment by the same practitioner for all 6 sessions. The healing touch practitioner will center his/her-self by bringing mind, body, and emotions into a quiet and focused state of mind. They will then assess the patient's energy field and implement healing touch techniques in the following order:

Chakra Connection Chakra Connection is a full body technique to open, connect, and balance the major and minor chakras and help clear the energy field. It promotes relaxation, reduces pain and anxiety and promotes general well-being and prevention.

Mind Clearing This HT technique is helpful in promoting mental clarity, peace, and calm. It facilitates deep relaxation, clear thinking, and promotes healthy sleep.

Chakra Spread. Chakra Spread is a gentle energy technique designed to open the chakras and produce a deep healing. It is helpful during life transitions to promote a deep sense of calm and peace - physically, emotionally, mentally, and spiritually.

No other forms of healing will be administered by the HT practitioner. The HT practitioner will use light touch to implement the healing touch techniques. Healing touch sessions will last approximately one hour and will occur two times per week for three weeks for a total of 6 sessions.

To complete the study, patients must receive all 6 sessions. For potential scheduling conflicts, exceptions will be made to accommodate patients for a maximum of 4 weeks.

Post-Intervention Assessment After 3 weeks, all participants in both groups will complete the following questionnaires: Dartmouth Quality of Life Index and SF-36 Health Survey.

All patients will enter the CR program as soon as the CR staff can schedule each patient.

Control Group When subjects in this group have completed their CR program they are offered a complementary one-time, one hour, healing touch treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Must have referral to Cardiac Rehab at the Scripps Center for Integrative Medicine.
2. Must have had a cardiac event which precede the CR referral.
3. Must be willing to come to the Scripps Center for Integrative Medicine twice a week for 3 weeks.
4. Must be able to understand English

Exclusion Criteria:

1. Patients under 18 years.
2. Unable to understand English

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2016-02; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with an improvement in stress and anxiety symptoms as measured by Dartmouth Quality of Life Index scores | 3 weeks
  Dartmouth Quality of Life Index questionnaires will be obtained at enrollment and after 3 weeks of HT (or no intervention for the control group).
Number of participants with an improvement in stress and anxiety symptoms as measured by SF-36 scores | 3 weeks
  SF-36 questionnaires will be obtained at enrollment and after 3 weeks of HT (or no intervention for the control group).

SECONDARY OUTCOMES:
Number of participants with an improvement of Metabolic Equivalent of Task (MET) | 3 months
  MET: Metabolic Equivalent of Task is measured at the start of Cardiac Rehab and at 3 months completion.
Number of participants with an improvement in BMI: Body Mass Index | 3 months
  BMI: Body Mass Index, which is measured at the start of Cardiac Rehab and at 3 months completion.
Number of participants with an improvement in stress and anxiety symptoms as measured by Dartmouth Quality of Life Index scores | 3 months
  Dartmouth Quality of Life Index scores will be obtained at the start of cardiac rehab and at completion.
Number of cardiac rehab sessions each participant attended will be recorded | 3 months
  To determine cardiac rehab attendance, study participants' number of sessions will be recorded. The program ends after 36 sessions (3 month). Not all participants complete all 36 sessions.
Number of participants with an improvement in stress and anxiety symptoms as measured by SF-36 scores | 3 months
  SF-36 scores will be obtained at the start of cardiac rehab and at completion.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Suhar, MD, Principal Investigator — Scripps Center for Integrative Medicine, Scripps Clinic
Locations (1):
- Scripps Center for Integrative Medicine, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No